CLINICAL TRIAL: NCT05947305
Title: Alternative Gingival De-Epithelialization Techniques: A Randomized Controlled Trial
Brief Title: Alternative Gingival De-Epithelialization Techniques
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Delta Dental Foundation (Other)
Responsible Party: Principal Investigator, Sandra Hyon Mi Stuhr, Clinical Assistant Professor of Dentistry, Periodontics and Oral Medicine, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HUM00231789
Record Dates: First submitted 2023-07-05; First posted 2023-07-17 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Recession, Gingival; Surgical Procedure, Unspecified; Graft Complication; Wound Heal
MeSH Terms: conditions — Gingival Recession | interventions — Lasers, Solid-State

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Surgical Blade (Placebo Comparator): A surgical blade will be used to de-epithelialize gum tissue during the subject's regularly scheduled dental surgery.
  Interventions: Procedure: Surgical Blade
- Mucotome (Experimental): A mucotome will be used to de-epithelialize gum tissue during the subject's regularly scheduled dental surgery.
  Interventions: Procedure: Mucotome
- Diamond Bur (Experimental): A diamond bur will be used to de-epithelialize gum tissue during the subject's regularly scheduled dental surgery.
  Interventions: Procedure: Diamond Bur
- Er:YAG Laser (Experimental): A dental laser will be used to de-epithelialize gum tissue during the subject's regularly scheduled dental surgery.
  Interventions: Procedure: Er:YAG Laser

INTERVENTIONS:
Procedure: Surgical Blade — Using a 15c blade to de-epithelialize the soft tissue extra-orally
  Arms: Surgical Blade
Procedure: Mucotome — Using Megagen Mucotome to de-epithelialize the soft tissue intra-orally
  Arms: Mucotome
Procedure: Diamond Bur — Using a surgical diamond bur to de-epithelialize the soft tissue intra-orally
  Arms: Diamond Bur
Procedure: Er:YAG Laser — Using an Er:YAG Laser to de-epithelialize the soft tissue intra-orally
  Arms: Er:YAG Laser

SUMMARY:
The goal of this clinical trial is to compare different de-epithelialization methods in patients undergoing soft tissue augmentation surgery. The main questions it aims to answer are:

• Which technique is superior for de-epithelialization in terms of remaining epithelium, wound healing of the donor site, and clinical outcomes?

DETAILED DESCRIPTION:
Participants will be randomly assigned to one of four surgical techniques during their surgical procedure and the wound site will be assessed on post-operative days 1, 7, 14, and 21.

Researchers will compare the use of mucotome, Er:YAG laser, surgical diamond bur, or blade to observe patterns of wound healing and assess if one method is superior in terms of removing the epithelium.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) Physical Status Classification I or II
* Subjects undergoing periodontal surgical procedures that involve harvesting of soft tissue samples, who have a treatment plan including the use or removal of keratinized mucosa or subepithelial connective tissue that will not require additional anesthesia for sample collection
* Adequate physical and mental health to undergo routine dental treatment
* Ability and willingness to follow instructions related to the study procedures

Exclusion Criteria:

* Poorly controlled diabetes, defined as HbA1c >/= 7.0
* Autoimmune or inflammatory conditions such as systemic lupus erythematous, rheumatoid arthritis.
* Pregnant women or nursing mothers, or unsure of pregnancy status (self-reported)
* Severe hematologic disorders, such as leukemia or hemophilia
* Subjects on anticoagulant or antiplatelet therapy
* Local or systemic infection that may interfere with healing
* Hepatic or renal diseases
* Currently under cancer treatment or within 18 months from completion of radio- or chemotherapy
* History of antibiotic or immunosuppressant use in the last 3 months
* Subjects on concomitant drug therapy for systemic conditions that may affect outcomes of the study
* Current smokers (CDC definition): heavy smokers: subjects who have smoked >10 cigarettes per day within 6 months of study onset, and have smoked >100 cigarettes in their lifetime

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-04-04 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Histomorphometric Comparison | After Day 0 (Baseline surgery)
  Histomorphometric evaluation of the relative proportion of epithelial tissue remnants (percentage) after de-epithelialization of the CTG

SECONDARY OUTCOMES:
Surgical Time | Day 0 (Baseline Surgery)
  Time spent removing the epithelium (in minutes)
Patient-reported outcome measures | Days 1, 7, 14, 21 (Post-operative) after surgery
  Patient-reported outcome measures regarding pain and discomfort after the procedure using a line scale (from no pain to worst pain imaginable), box scale (ranging from 0-10 with 0 being no pain and 10 being worst pain imaginable), and a verbal rating scale (no pain, slightly painful, moderately painful, very painful, extremely painful). The number of analgesics (along with dosage) taken during the post-operative period will be recorded.
Wound healing | Days 1, 7, 14, 21 (Post-operative) after surgery
  Wound healing comparisons using a clinical healing index (CHI) developed by Pippi et al 2015 will be completed. The possible total score is 7 (ideal score demonstrating ideal healing = 0), with scores for each section being dichotomous (0 or 1). Parameters related to clinical inspection include: mucosal color, granulation tissue, epithelialization degree, and swelling. Palpation parameters include bleeding, pain, and suppuration.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Stuhr, DMD, MS, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan School of Dentistry, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zucchelli G, Tavelli L, McGuire MK, Rasperini G, Feinberg SE, Wang HL, Giannobile WV. Autogenous soft tissue grafting for periodontal and peri-implant plastic surgical reconstruction. J Periodontol. 2020 Jan;91(1):9-16. doi: 10.1002/JPER.19-0350. Epub 2019 Oct 6. PMID 31461778
- [Background] Chambrone L, Chambrone D, Pustiglioni FE, Chambrone LA, Lima LA. Can subepithelial connective tissue grafts be considered the gold standard procedure in the treatment of Miller Class I and II recession-type defects? J Dent. 2008 Sep;36(9):659-71. doi: 10.1016/j.jdent.2008.05.007. Epub 2008 Jun 26. PMID 18584934
- [Background] Zuhr O, Baumer D, Hurzeler M. The addition of soft tissue replacement grafts in plastic periodontal and implant surgery: critical elements in design and execution. J Clin Periodontol. 2014 Apr;41 Suppl 15:S123-42. doi: 10.1111/jcpe.12185. PMID 24640997
- [Background] Dellavia C, Ricci G, Pettinari L, Allievi C, Grizzi F, Gagliano N. Human palatal and tuberosity mucosa as donor sites for ridge augmentation. Int J Periodontics Restorative Dent. 2014 Mar-Apr;34(2):179-86. doi: 10.11607/prd.1929. PMID 24600654
- [Background] Sanz-Martin I, Rojo E, Maldonado E, Stroppa G, Nart J, Sanz M. Structural and histological differences between connective tissue grafts harvested from the lateral palatal mucosa or from the tuberosity area. Clin Oral Investig. 2019 Feb;23(2):957-964. doi: 10.1007/s00784-018-2516-9. Epub 2018 Jun 18. PMID 29915931
- [Background] Tavelli L, Barootchi S, Ravida A, Oh TJ, Wang HL. What Is the Safety Zone for Palatal Soft Tissue Graft Harvesting Based on the Locations of the Greater Palatine Artery and Foramen? A Systematic Review. J Oral Maxillofac Surg. 2019 Feb;77(2):271.e1-271.e9. doi: 10.1016/j.joms.2018.10.002. Epub 2018 Oct 11. PMID 30395825
- [Background] Edel A. Clinical evaluation of free connective tissue grafts used to increase the width of keratinised gingiva. J Clin Periodontol. 1974;1(4):185-96. doi: 10.1111/j.1600-051x.1974.tb01257.x. No abstract available. PMID 4533490
- [Background] Langer B, Langer L. Subepithelial connective tissue graft technique for root coverage. J Periodontol. 1985 Dec;56(12):715-20. doi: 10.1902/jop.1985.56.12.715. PMID 3866056
- [Background] Harris RJ. The connective tissue and partial thickness double pedicle graft: a predictable method of obtaining root coverage. J Periodontol. 1992 May;63(5):477-86. doi: 10.1902/jop.1992.63.5.477. PMID 1527693
- [Background] Carranza N, Rojas MA. Bilaminar Palatal Connective Tissue Grafts Obtained With the Modified Double Blade Harvesting Technique: Technical Description and Case Series. Clin Adv Periodontics. 2020 Dec;10(4):186-194. doi: 10.1002/cap.10124. Epub 2020 Sep 20. PMID 32862553
- [Background] Wei PC, Geivelis M. A gingival cul-de-sac following a root coverage procedure with a subepithelial connective tissue submerged graft. J Periodontol. 2003 Sep;74(9):1376-80. doi: 10.1902/jop.2003.74.9.1376. PMID 14584873
- [Background] El-Kholey KE. Efficacy and safety of a diode laser in second-stage implant surgery: a comparative study. Int J Oral Maxillofac Surg. 2014 May;43(5):633-8. doi: 10.1016/j.ijom.2013.10.003. Epub 2013 Nov 7. PMID 24210453
- [Result] Bosco AF, Bosco JM. An alternative technique to the harvesting of a connective tissue graft from a thin palate: enhanced wound healing. Int J Periodontics Restorative Dent. 2007 Apr;27(2):133-9. PMID 17514885
- [Result] Zucchelli G, Amore C, Sforza NM, Montebugnoli L, De Sanctis M. Bilaminar techniques for the treatment of recession-type defects. A comparative clinical study. J Clin Periodontol. 2003 Oct;30(10):862-70. doi: 10.1034/j.1600-051x.2003.00397.x. PMID 14710766
- [Result] Zucchelli G, Mele M, Stefanini M, Mazzotti C, Marzadori M, Montebugnoli L, de Sanctis M. Patient morbidity and root coverage outcome after subepithelial connective tissue and de-epithelialized grafts: a comparative randomized-controlled clinical trial. J Clin Periodontol. 2010 Aug 1;37(8):728-38. doi: 10.1111/j.1600-051X.2010.01550.x. Epub 2010 Jun 24. PMID 20590963
- [Result] Tavelli L, Ravida A, Lin GH, Del Amo FS, Tattan M, Wang HL. Comparison between Subepithelial Connective Tissue Graft and De-epithelialized Gingival Graft: A systematic review and a meta-analysis. J Int Acad Periodontol. 2019 Apr 1;21(2):82-96. PMID 31522155